CLINICAL TRIAL: NCT05821608
Title: Evaluating the Impact of 'Heads up' Messages on Call Pick-up Rates
Brief Title: Heads up Messages to Increase Call Pick-up Rates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Carnegie Mellon University (Other)
Responsible Party: Principal Investigator, George Loewenstein, Professor, Carnegie Mellon University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: HEADSUP2
Record Dates: First submitted 2023-04-07; First posted 2023-04-20 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Various: Health Insurance Members That Could Benefit From Being Connected to a Specialist, e.g., Orthopedic Doctor to Treat Back Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not know treatment status but callers and investigators will not be blinded to treatment status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Participants will not receive a message before a nurse tries to contact them via a phone call.
- Heads Up Message 1 (Experimental): Participants will receive a message before a nurse tries to contact them via a phone call with the following text:
  Hi @{account_firstname}, this is @{input_MEGname} at @{account_product_group}. Just a heads up, I'm calling in the next hour about your health care. Text help or stop. Msg&DataRatesMayApply
  Interventions: Other: Message variation 1
- Heads Up Message 2 (Experimental): Participants will receive a message before a nurse tries to contact them via a phone call with the following text:
  Hi @{account_firstname}, this is @{input_MEGname} at @{account_product_group}. Just a heads up, I'm calling in the next hour about your health care. Text HELP for Help and Text STOP to Stop. (Note: replying STOP will stop all further texts from @{account_product_group}). Msg&DataRatesMayApply
  Interventions: Other: Message variation 2

INTERVENTIONS:
Other: Message variation 1 — Message before call letting member know they will be called (variation 1)
  Arms: Heads Up Message 1
Other: Message variation 2 — Message before call letting member know they will be called (variation 2)
  Arms: Heads Up Message 2

SUMMARY:
The study aims to investigate whether notifying health insurance members about an upcoming call can increase their pick-up rates. The study will randomize participants into three groups: control group (no message), treatment group 1 (message variation 1), and treatment group 2 (message variation 2). The primary outcome of interest is the call pick-up rate, and the study will also examine the message opt-out rates for the two different messages.

ELIGIBILITY:
Inclusion Criteria:

* The study will include members enrolled in the health insurers' Relay Texting system due to receive an outreach call during the study timeframe.
* Enrollment in the study will end when we meet our enrollment target (N=2000)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants who pick up the phone call | The time between the second and first call attempt may vary but will be less than 10 days.
  All members in the study will receive two call attempts. The outcome will be positive if the calling nurse gets through to the member on either the first or second call attempt, and negative otherwise.

SECONDARY OUTCOMES:
Percentage of participants who opt out of future text messages | We will consider a member as opted out if they opt out of messages within 24 hours of receiving a message as part of the study.
  We will measure whether members opt out of receiving any text messages from the insurer in response to the heads up messages.

IPD SHARING:
Plan to Share IPD: No